CLINICAL TRIAL: NCT04929704
Title: Diagnostic Yield and Influence on Length of Stay of Brain Computed Tomography for Elderly Patients With Altered Mental Status in an Emergency Setting
Acronym: DISCUSS-CT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DISCUSS-CT
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-04

CONDITIONS: Altered Mental Status
Keywords: elderly patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The confusional syndrome is defined by the acute or subacute onset of a deficit syndrome (temporo-spatial disorientation, memory and concentration disorders, abnormal behavior, impairment of intellectual efficiency, fluctuation of disorders with an increase in the evening) that may be associated with a productive syndrome (visual or auditory hallucinations, delusional elements) (French College of Neurology). It is a frequent, serious and costly problem in hospitalized patients and in emergency rooms.

Its prevalence is between 10 and 31% of cases in emergency rooms and concerns up to one out of two elderly patients during a hospitalization. The potential morbidity and mortality of the confusional syndrome is due in part to the difficulty of identifying and treating rapidly the triggering and aggravating factors that are often interrelated in the elderly. Most often, these are drug effects, metabolic disorders, infections, consequences of prolonged immobilization or physical restraint. The lack of rapid treatment of these causes increases the risk of medium and long-term cognitive problems.

Because of the aging population, this is an increasingly expensive problem. In 2012, the World Health Organization Regional Office for Europe study conducted in 18 European countries combined estimated its cost at $182 billion per year. The management of confusional syndrome in the elderly is now a major public health issue. It is a targeted indicator of the safety and quality of care for the elderly.

DETAILED DESCRIPTION:
However, in the majority of situations, an appropriate history, an analysis of the patient's treatments, a rigorous physical examination, and a blood biology examination are sufficient to quickly identify and treat the cause(s) of the confusional syndrome. In the practice of emergency departments, a brain scan without injection of contrast medium is nevertheless frequently prescribed for an elderly person presenting a recent alteration of his cognitive functions. One explanation is that clinical signs suggestive of intracranial lesion may be more difficult to detect in frail elderly patients with a significant history, in the same way as those of sepsis for example. On the other hand, an alteration of the cognitive function without any known antecedents for the patient, probably leads emergency physicians to suspect too frequently a central neurological cause. However, the cause is most often of extracerebral origin.

At Paris Saint Joseph Hospital, the number of emergency room visits increased by 4% between 2018 and 2019. The Emergency Department is the second largest emergency department in Ile de France in terms of attendance of a geriatric patient base (20% of patients seen). These observations prompt an urban emergency department like ours to evaluate the relevance and quality of our geriatric emergency medicine practices.

In the literature, several American studies, mostly monocentric and retrospective, have examined the diagnostic utility of brain scans in elderly patients with confusional syndromes during their observation in the emergency department. The discovery of a scannographic abnormality explaining the symptomatology occurred in 10 to 39% of cases depending on the series. The patient cohorts differed in terms of age and clinical presentation. Some were predominantly composed of patients with a focal neurological sign associated with confusion, others exclusively of patients with head trauma. We did not find any study that specifically evaluated the diagnostic contribution of an emergency brain scan in the elderly patient ≥ 75 years of age with isolated confusion, i.e., in the absence of a neurological localizing sign and in the absence of a head injury under antiplatelet therapy (AAP) and/or anticoagulant therapy, for which the indication of brain imaging is not debatable. One study evaluated the diagnostic yield of brain scans in the emergency department in adult patients with an acute delirious episode. However, it was more about exploring a first psychiatric episode in rather young patients. This problem appears interesting in the confused elderly subject because the realization of a CT scan is time-consuming, expensive, and irradiating. It has an impact on the length of stay in the emergency department, the prolongation of which is itself a source of a confusional episode, with its share of complications: fall, agitation, disorientation, mechanical restraint, inappropriate use of benzodiazepines and neuroleptics, for example.

Given the ageing of the population, the morbidity of confusional episodes in the elderly in the absence of rapid adapted treatment, and the frequent saturation of emergency departments, it is useful to know the real diagnostic yield of the brain scan performed for an isolated confusional syndrome observed in the elderly in the emergency department. At the same time, in France, targeted studies have highlighted an unregulated growth in the prescription of certain medical imaging procedures. Possible reasons for this include the practice of defensive medicine by extension of the precautionary principle, and the high expectations of patients, their relatives, or treating physicians, who may exert pressure to prescribe. Finally, acting also under the pressure of time management, where the clinical time spent with each patient tends to be reduced, it is paradoxical that the prescription of brain imaging examinations has increased in the emergency department in recent years. Determining the organizational impact on the duration of care would allow us to meet a quality of care objective.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ⩾ 75 years who had a brain scan without contrast injection in the emergency department due to isolated confusional syndrome between January 1, 2019 and December 31, 2019.
* French-speaking patient

Exclusion Criteria:

* Patient with concomitant localizing neurological signs of confusional syndrome: abnormalities of the cranial pairs, unusual headaches, meningeal syndrome, cerebellar syndrome, systematized sensory or motor deficit, vestibular syndrome, Glasgow Coma Scale score ≤ 8.
* Patient who has had a head injury and is taking a long-term antiplatelet and/or anticoagulant therapy.
* Patient objecting to the use of their data for this research.
* Patient deprived of liberty
* Patient under court protection

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient aged ⩾ 75 years who had a brain scan without contrast injection in the emergency department due to isolated confusional syndrome between January 1, 2019 and December 31, 2019.
Sampling Method: Non-Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-07-11 (Actual); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Determine the diagnostic yield of brain scans without contrast injection for patients aged ≥ 75 years with isolated confusional syndrome (proportion of scans explaining symptomatology) | Day 1
  Evidence of a recent intracranial abnormality compatible with the patient's symptomatology (isolated confusional syndrome)

SECONDARY OUTCOMES:
To determine the impact of performing an injection-free brain scan to patients aged ≥ 75 years with isolated confusional syndrome on the duration of their emergency department management. | Day 1
  Increase in the length of time spent in the emergency room related to the performance of the brain scan (time between the time the brain scan is ordered and the time it is interpreted).
Identify the anamnestic, clinical, and biological variables available in the emergency department associated with the discovery of an intracranial process on CT explaining the clinical picture. | Day 1
  Anamnestic, clinical, and biological parameters available in the emergency department statistically associated with the occurrence of the primary outcome.
To determine the main etiology of the confusional syndrome in patients whose CT scan did not find an acute abnormality explaining the symptomatology. | Day 1
  Main causes of confusional syndromes not explained by an acute intracranial anomaly on CT.
Determine the impact of the CT scan result on the patient's initial medical management strategy (first 24 hours). | Day 1
  Modification of the diagnostic approach (addition of a complementary examination such as brain MRI or EEG) or therapeutic approach (discontinuation or addition of a drug treatment, surgical or radio-interventional management), or filiarization (hospitalization in neurology, neurovascular continuous care unit, neurosurgery, or intensive care unit)

CONTACTS AND LOCATIONS:
Overall Officials: Camille GERLIER, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France